CLINICAL TRIAL: NCT01474694
Title: Accuracy Assessment for Computer-assisted Surgical Interventions of the Liver: A Prospective, Non Randomized Study
Brief Title: Accuracy Assessment for Computer-assisted Surgical Interventions of the Liver
Acronym: CALS
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr.med. Vanessa Banz/ Prof. Dr. med.Daniel Candinas, Bern University Hospital
Other Study IDs: 063/11; Eureka 6201/5/Ae
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Adult Liver Cancer
Keywords: prospective study; multicenter trial; analysis, computer assisted image; CE marked; medical devices; catheter ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Abdominal surgery — The patient is placed in a supine position and standard laparotomy (either via subcostal, midline or inverted hockey-stick incision) is performed. After mobilization of the liver, surgical swabs are packed around the organ to prevent unnecessary movement of the liver during the acquisition of the landmarks and the subsequent surgical procedure

SUMMARY:
Preoperative image-guided data correlates with the actual intraoperative reality. Computer-assisted preoperative planning combined with intraoperative mapping of even very small lesions allows for improved accuracy during complete oncological resection / ablation. In the short- and long-term this possibly results in better patient outcome.

DETAILED DESCRIPTION:
Background

The aim of this study is to analyze the available accuracy of a computer-assisted approach to liver surgery and microwave ablation. The term 'computer-assisted' refers to 1) using 3D models of patient anatomy for extended orientation during the planning of the intervention and 2) using an image guidance system (similar to a GPS in a car) that allows for precise targeting of desired anatomical structures (e.g. intrahepatic tumor, bile ducts / vasculature) in the setting of successfully treating liver malignancies. Furthermore, we would like to demonstrate, that image guided open liver surgery is technically feasible, whenever the correlation between preoperative image-guided data and the intraoperative setting can be achieved with a known accuracy.

Eventually, this technology, like in other surgical domains, will lead to successively implemented technical guiding functionalities that could potentially improve patient outcome.

Objective

To date, first systems (CE marked medical devices) are available that have been specifically developed for image-guided open liver surgery. The systems tracks positions of surgical instruments in or near the target organs and visualizes the instruments position in correlation to patients medical image data (i.e. 3D-CT) on the computer screen. Surgeons benefit from a view to a virtual scene (on a computer screen) in which CT images, together with models of the vascular structures, tumors and organ boundaries, are intuitively visible. The surgeon can see the moving instrument, just like the movement of a car can be seen in a GPS system

Methods

In patients requiring extensive surgery (eg. extended right hemihepatectomy), accurate calculations of the remaining liver volume are essential to avoid postoperative liver failure with potentially serious postoperative complications or even death, resulting from an inadequate remaining liver volume (ie "small-for-size syndrome"). In high-risk liver resections, use of computer programs, such as MeVis (MeVis Medical Solutions Inc.), provide the surgeon with accurate preoperative information, allowing him / her to judge the feasibility of the planned surgical resection based on preoperative liver volume analysis and evaluation of the planned resection line in relation to essential structures (ie. major vessels / bile ducts).

ELIGIBILITY:
Inclusion Criteria:

* 1.Written informed consent
* 2.Male patients and non-pregnant, non-lactating females aged ≥18 years of age (negative serum/urine pregnancy test result at screening)
* 3.Patients must be candidates for surgical liver resection and/or MWA (at least one anatomical segment) of primary or metastatic liver cancer. The liver tumors must be present on preoperative imaging study (CT and/or MRI).

Exclusion Criteria

* 1.Any condition which, in the judgment of the clinical investigator or his designee, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
* 2.A mental condition rendering the patient unable to provide informed consent.
* 3.Patients with hereditary hematological / coagulation disorders unrelated to their liver disease or cirrhosis of the liver classified as Child's B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that are still considered unresectable at the time point of presentation
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
TRE, measuring the error in the prediction of a surgical target location when using the navigation system. | 12 months

SECONDARY OUTCOMES:
1.Identification of suitable landmarks for registration | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Banz, Dr. med., Principal Investigator — Bern University Hospital; Daniel Candinas, Prof. Dr. med., Principal Investigator — Bern University Hospital
Locations (1):
- Dep. of visceral and Transplant Surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Peterhans M, vom Berg A, Dagon B, Inderbitzin D, Baur C, Candinas D, Weber S. A navigation system for open liver surgery: design, workflow and first clinical applications. Int J Med Robot. 2011 Mar;7(1):7-16. doi: 10.1002/rcs.360. Epub 2010 Oct 29. PMID 21341357
- [Background] Gavaghan KA, Peterhans M, Oliveira-Santos T, Weber S. A portable image overlay projection device for computer-aided open liver surgery. IEEE Trans Biomed Eng. 2011 Jun;58(6):1855-64. doi: 10.1109/TBME.2011.2126572. Epub 2011 Mar 14. PMID 21411401